CLINICAL TRIAL: NCT03376061
Title: DEPOSITION: Pilot Study Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery
Brief Title: Decreasing Postoperative Blood Loss by Topical vs. Intravenous Tranexamic Acid in Open Cardiac Surgery
Acronym: DEPOSITION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEPOSITION 1.0 2017-07-28
Record Dates: First submitted 2017-11-17; First posted 2017-12-18 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Bleeding; Surgical Blood Loss
Keywords: Tranexamic Acid; Cardiac surgery
MeSH Terms: conditions — Hemorrhage; Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Tranexamic Acid intravenous + Placebo topical versus Placebo intravenous + Tranexamic Acid topical
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy will prepare 1 syringe of 50 ml of topical TA (5 g) or placebo. They will also prepare for the same patient 2 syringes of 50 ml (5 g) for intravenous (i.v.) injection or placebo. TA is similar in all aspects to normal saline. Blinding of both teams will be easy. The syringes will be prepared and randomized in pharmacy before the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TA Topical (Active Comparator): 1 syringe of 50ml of topical Tranexamic Acid (5g) or placebo. The topical will be poured into the pericardial mediastinal cavities in 2 equal doses, 25ml when the pt comes off-pump and the other 25ml before sternotomy is closed.
  Interventions: Drug: Tranexamic Acid
- TA Intravenous (Active Comparator): 2 syringes of 50ml (5mg) Tranexamic Acid for intravenous injection or placebo.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic Acid is a medication used to treat or prevent excessive blood loss from major trauma, post partum, surgery, tooth removal, nose bleeds, and heavy menstruation.
  Other Names: Cyklokapron

SUMMARY:
The aim is to conduct a double-blinded single-centre randomized controlled clinical trial of application of topical dose of tranexamic acid (TA) versus the usual intravenous TA in patients undergoing cardiac surgery at the Hamilton General Hospital. This pilot study will assess the feasibility to perform a large randomized international trial exploring this objective.

DETAILED DESCRIPTION:
Postoperative bleeding related to open cardiac surgery increases the rates of complications and mortality. It results from the blood thinners that are needed for use. Intravenous tranexamic acid (TA) has become a mainstay in cardiac surgical procedures for decreasing bleeding and minimizing transfusion requirements. Although intravenous TA is usually well tolerated, there is a well-known risk (1 to 4%) of postoperative seizures. This is due to the similarity between TA and the brain tissues. The aim is to eliminate the risk of seizures but to maintain the protection against bleeding. When TA is used directly on the tissues (topically) for other type of surgeries (joints), TA is effective to reduce blood loss and transfusions. The aim is to prove that direct application of TA on the heart can eliminate postoperative seizures and reduce the amount of blood transfusions in patients who have cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >= 18 years old
* Undergoing cardiac surgical procedure with the use of cardiopulmonary bypass and median sternotomy
* Provide written informed consent

Exclusion Criteria:

* Poor (English) language comprehension
* Minimally invasive valve surgery
* Off-pump procedures
* Emergency operations
* Known history of increased bleeding disorder
* Thromboembolic disease
* Allergy to tranexamic acid
* Severe renal impairment (eGFR <30 mL/min/1.73m2 )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD MHSc, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kucuk O, Kwaan HC, Frederickson J, Wade L, Green D. Increased fibrinolytic activity in patients undergoing cardiopulmonary bypass operation. Am J Hematol. 1986 Nov;23(3):223-9. doi: 10.1002/ajh.2830230306. PMID 3766524
- [Background] Harker LA, Malpass TW, Branson HE, Hessel EA 2nd, Slichter SJ. Mechanism of abnormal bleeding in patients undergoing cardiopulmonary bypass: acquired transient platelet dysfunction associated with selective alpha-granule release. Blood. 1980 Nov;56(5):824-34. No abstract available. PMID 6448643
- [Background] Despotis GJ, Santoro SA, Spitznagel E, Kater KM, Cox JL, Barnes P, Lappas DG. Prospective evaluation and clinical utility of on-site monitoring of coagulation in patients undergoing cardiac operation. J Thorac Cardiovasc Surg. 1994 Jan;107(1):271-9. PMID 8283896
- [Background] Lemmer JH Jr, Stanford W, Bonney SL, Breen JF, Chomka EV, Eldredge WJ, Holt WW, Karp RB, Laub GW, Lipton MJ, et al. Aprotinin for coronary bypass operations: efficacy, safety, and influence on early saphenous vein graft patency. A multicenter, randomized, double-blind, placebo-controlled study. J Thorac Cardiovasc Surg. 1994 Feb;107(2):543-51; discussion 551-3. PMID 7508070
- [Background] Santos AT, Kalil RA, Bauemann C, Pereira JB, Nesralla IA. A randomized, double-blind, and placebo-controlled study with tranexamic acid of bleeding and fibrinolytic activity after primary coronary artery bypass grafting. Braz J Med Biol Res. 2006 Jan;39(1):63-9. doi: 10.1590/s0100-879x2006000100007. Epub 2005 Dec 15. PMID 16400465
- [Background] Pleym H, Stenseth R, Wahba A, Bjella L, Karevold A, Dale O. Single-dose tranexamic acid reduces postoperative bleeding after coronary surgery in patients treated with aspirin until surgery. Anesth Analg. 2003 Apr;96(4):923-928. doi: 10.1213/01.ANE.0000054001.37346.03. PMID 12651635
- [Background] Myles PS, Smith JA, Forbes A, Silbert B, Jayarajah M, Painter T, Cooper DJ, Marasco S, McNeil J, Bussieres JS, McGuinness S, Byrne K, Chan MT, Landoni G, Wallace S; ATACAS Investigators of the ANZCA Clinical Trials Network. Tranexamic Acid in Patients Undergoing Coronary-Artery Surgery. N Engl J Med. 2017 Jan 12;376(2):136-148. doi: 10.1056/NEJMoa1606424. Epub 2016 Oct 23. PMID 27774838
- [Background] Martin K, Wiesner G, Breuer T, Lange R, Tassani P. The risks of aprotinin and tranexamic acid in cardiac surgery: a one-year follow-up of 1188 consecutive patients. Anesth Analg. 2008 Dec;107(6):1783-90. doi: 10.1213/ane.0b013e318184bc20. PMID 19020118
- [Background] Kalavrouziotis D, Voisine P, Mohammadi S, Dionne S, Dagenais F. High-dose tranexamic acid is an independent predictor of early seizure after cardiopulmonary bypass. Ann Thorac Surg. 2012 Jan;93(1):148-54. doi: 10.1016/j.athoracsur.2011.07.085. Epub 2011 Nov 4. PMID 22054656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2017 and April 2018 a total of 97 patients were randomized to the topical (n = 49) and intravenous (n = 48) groups.
Groups:
- Topical TxA (Intervention): 50 mL of topical tranexamic acid (equivalent to 5 g TxA) poured into the pericardial and mediastinal cavities in 2 equal doses: 25 mL when the patient comes off-pump and the remaining 25 mL before sternotomy closure. In addition, patients received intravenous placebo (saline) administered as per anesthetist standard of care.
- Intravenous TxA (Control): Up to 100 mL of intravenous tranexamic acid (equivalent to 10 g TxA) administered as per anesthetist standard of care. In addition, patients will receive topical placebo (saline) poured into the pericardial and mediastinal cavities in 2 equal doses: 25 mL when the patient comes off-pump and the remaining 25 mL before sternotomy closure.
Period: Overall Study
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Started | 49 | 48
Completed | 49 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Topical TxA (Intervention): 50 mL of topical tranexamic acid (equivalent to 5 g TxA) poured into the pericardial and mediastinal cavities in 2 equal doses: 25 mL when the patient comes off-pump and the remaining 25 mL before sternotomy closure. In addition, patients will receive intravenous placebo (saline) administered as per anesthetist standard of care.
- Total: Total of all reporting groups
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control) | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (9.4) | 67.8 (9.2) | 67.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 44 | 42 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 46 | 46 | 92
  Hispanic/Latino | 0 | 2 | 2
  Southeast Asian/Malaysian | 1 | 0 | 1
  Aboriginal/Native Persons | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 49 | 48 | 97
Diabetes mellitus [Count of Participants; unit: Participants] | 17 | 21 | 38
Stroke [Count of Participants; unit: Participants] | 3 | 3 | 6
Transient ischemic attack [Count of Participants; unit: Participants] | 2 | 2 | 4
Carotid endarterectomy/stent [Count of Participants; unit: Participants] | 3 | 1 | 4
History of seizures [Count of Participants; unit: Participants] | 1 | 0 | 1
New oral anticoagulants (NOAC) [Count of Participants; unit: Participants] | 3 | 4 | 7
Aspirin [Count of Participants; unit: Participants] | 38 | 42 | 80
Clopidogrel (Plavix) [Count of Participants; unit: Participants] | 12 | 7 | 19
Ticagrelor [Count of Participants; unit: Participants] | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Median Volume of Mediastinal Fluid Collected From Participants
Description: Cumulative volume (mL) of fluid collected from mediastinal drainage tubes 24 hours after the surgical procedure
Time Frame: Fluid collected in the first 24 hours after the surgical procedure
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 49 | 48
mL | 500 [350 to 750] | 540 [420 to 700]

2. Secondary Outcome: Number of Participants With Seizures
Description: Patients experiencing a post-operative seizure
Time Frame: Patients will be followed post-operatively until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 49 | 48
Participants | 0 | 1

3. Secondary Outcome: Number of Participants With Mortality
Description: The occurrence of death due to any cause
Time Frame: Patients will be followed post-operatively until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 49 | 48
Participants | 1 | 1

4. Secondary Outcome: Number of Participants With RBC Transfusion
Description: Patients requiring a red blood cell transfusion
Time Frame: Intra-operative and post-operative RBC transfusions
Measure: Count of Participants; unit: Participants
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 49 | 48
Participants | 19 | 23

5. Secondary Outcome: Number of Participants With Re-operation for Bleeding or Tamponade
Description: Occurrence of re-operation for the purpose of bleeding or cardiac tamponade
Time Frame: Patients will be followed post-operatively until hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 49 | 48
Participants | 0 | 1

6. Secondary Outcome: Median Number of Hours Participants Spent in ICU
Description: Number of hours participants spent in the intensive care unit (ICU)
Time Frame: Number of hours spent in ICU from arrival to exit (collected at the Post-Operative Visit).
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 49 | 48
hours | 23 [19 to 45] | 26 [22 to 53]

7. Secondary Outcome: Mean Concentration of TxA in Plasma Collected From Participants
Description: Plasma TxA concentrations measured from blood samples taken upon arrival in the ICU
Time Frame: on arrival in ICU within 3 hours
Population: 4 patients from the topical TxA group and 3 patients from the intravenous TxA group were excluded because they either did not receive a TxA dose or received an incomplete TxA dose.
Measure: Mean (Standard Deviation); unit: microgram per milliliter per kilogram
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
Number analyzed (Participants) | 45 | 45
microgram per milliliter per kilogram | 0.58 (0.41) | 1.10 (0.52)

ADVERSE EVENTS:
Time Frame: 30 days post-operatively
Arm/Group | Topical TxA (Intervention) | Intravenous TxA (Control)
All-Cause Mortality (participants affected / at risk) | 1/49 | 1/48
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48
Other Adverse Events (participants affected / at risk) | 0/49 | 0/48

LIMITATIONS AND CAVEATS:
Due to the small sample size (N<100 patients) the DEPOSITION pilot trial is not sufficiently powered to detect statistically significant differences between topical and intravenous TxA groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT03376061/Prot_SAP_000.pdf